CLINICAL TRIAL: NCT01633203
Title: Prospective Observational Study of Patients With Locally Advanced Gastric Cancer Treated With Perioperative Chemotherapy and Surgery
Brief Title: Observational Study of Perioperative Chemotherapy in Gastric Cancer
Acronym: PRECISO
Status: Completed | Type: Observational
Sponsor: Grupo Oncologico Cooperativo Chileno de Investigation (Network)
Responsible Party: Sponsor
Other Study IDs: GOCCHI 2009-01
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; combination chemotherapy; HER-2 gene; quality of life
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Cisplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- locally advanced gastric cancer: Patients with resectable, locally advanced cT3-4 and/or N+ gastric carcinoma treated with 3 perioperative epirubicin cisplatin capecitabine polychemotherapy
  Interventions: Drug: epirubicin + cisplatin + capecitabine polychemotherapy

INTERVENTIONS:
Drug: epirubicin + cisplatin + capecitabine polychemotherapy — EPIRUBICIN (LKM)at a dose of 50 mg/m2 over 15 minutes is administered every 21 days.
  CISPLATIN (LKM) at a dose of 60 mg/m2 over 4 hours is administered every 21 days. Patients must receive standardized hydration per protocol.
  CAPECITABINE (Xeloda®) at a dose of 625 mg/m2 BID (i.e. 1250 mg/m2/day) 30 minutes after meals from day 1 to day 21 of every cycle of chemotherapy.
  Antiemetic therapy:
  * Dexamethasone 8 mg IV and Ondansetron (LKM) 8 mg IV o Granisetron (Kytril®) prior to chemotherapy
  * Rescue Ondansetron (LKM) 8 mg IV will be given during 24-hour hospitalization in case of emesis
  * Symptomatic antiemetic therapy with thiethylperazine will be prescribed.
  Loperamide will be prescribed in case of diarrhea.

SUMMARY:
This study will assess the efficacy and toxicity of perioperative chemotherapy with Epirubicin + Cisplatin + Capecitabine (ECX) in routine clinical practice in a network of public hospitals in Santiago, Chile.

DETAILED DESCRIPTION:
Chile belongs to the countries with a high mortality rate due to gastric cancer, and this disease is the most frequent cause of cancer death in Chile. Despite of adequate surgery, survival rates are disappointing, with less than 60% of patients for all stages achieving to be alive at 5 years. This is due to the fact that frequently gastric cancer is diagnosed at an advanced stage. For locally advanced gastric cancer a multimodality treatment is recommended, with the alternatives of surgery followed by chemotherapy (asian approach), surgery followed by chemoradiation (US approach) and perioperative chemotherapy (european approach). These three strategies are valid standard treatment options and have shown to improve overall survival in stage IB to IVA gastric cancer.

Perioperative chemotherapy administered pre- and postoperatively, has shown to downstage the tumor, increase curative resection, progression free and overall survival.

For patients with potentially resectable gastric cancer staged T2 or higher or cN+, NCCN Guidelines recommend perioperative chemotherapy (category1). Chilean guidelines for gastric cancer state the alternative of perioperative chemotherapy, however this approach has not been used widely in public hospitals because lack of financial support.

Some gastric cancers overexpress HER2, and this subset of patients benefit from targeted therapy at an advanced stage. The proportions of patients with these molecular characteristics vary widely depending of the geographic area. The chilean population has been investigated in small series, but the incidence of HER2 positive gastric cancer is not known. We therefore plan to measure HER2 expression in all participating patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive carcinoma
* Age > 18 years.
* ECOG performance status 0 or 1.
* Hemoglobin > 9 g/dL
* Absolute neutrophil count > 1.5 x 109/L
* Platelet count > 100 x 109/L
* Creatinine < 1.5 ULN
* Creatinine clearance > 60 mL/min
* Serum bilirubin < 1.5 x ULN
* AST < 2.5 x ULN
* Women of child bearing potential: must agree to use an effective contraceptive method.
* Signed informed consent.

Exclusion Criteria:

* ECOG > 2.
* Pre-existing diarrhea uncontrolled with supportive care.
* Inability to swallow Xeloda tablets.
* History of mild-to-moderate renal insufficiency (creatinine clearance < 45 mL/min).
* Signs or symptoms of clinically significant hepatic dysfunction (bilirubin > 1.5 ULN, FA > 2.5 ULN, albumin < 2,5 g/dL).
* Significant cardiac dysfunction (LVEF < LLN)
* Presence of distant metastasis, including clinical signs of peritoneal carcinomatosis
* Symptomatic gastric retention or severe dysphagia with a caloric intake of < 1500 kcal/day
* Histology of lymphoma, GIST or neuroendocrine tumor
* Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile or they must agree to use an effective method of contraception.
* Any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include congestive heart failure of Class III or IV of the NYHA classification, infection requiring parental or oral treatment, any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current diagnosis of T3-4 and/or N+ M0 (according to staging system of the American Joint Committee on Cancer 2002) resectable gastric cancer. The resectability has to be confirmed by a surgical oncologist and/or Oncological Committee.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Rate of downstaging | through study completion, an average of 3 months
  To determine the rate of downstaging of locally advanced cT3-4 and/or N+ gastric carcinomas after 3 cycles of preoperative chemotherapy with ECX

SECONDARY OUTCOMES:
Rate of adverse events | through study completion, an average of 6 months
  Rate and description of adverse events
Clinical response after three cycles of preoperative ECX | through study completion, an average of 6 months
  Clinical response based on RECIST criteria
To evaluate the surgical morbidity after three cycles of preoperative CT | through study completion, an average of 1 year
  Hospital stay duration
To evaluate the surgical mortality after three cycles of preoperative CT | through study completion, an average of 1 year
  30 days postoperative mortality rate
progression free survival | through study completion, an average of 2 years
  To evaluate the 3 year progression free survival
overall survival | through study completion, an average of 3 years
  To evaluate the 5 year overall survival (OS) of patients treated with perioperative CT
compliance with the planned postoperative therapy | through study completion, an average of 1 year
  To evaluate the rate of start and completion of postoperative treatment
EORTC QLQ-C30 after neoadjuvant chemotherapy and surgery | through study completion, an average of 2 years
  To evaluate quality of life through patient reported outcomes of patients treated with perioperative chemotherapy
EORTC QLQ-STO 22 after neoadjuvant chemotherapy and surgery | through study completion, an average of 2 years
  To evaluate patient reported specific symptoms of patients treated with perioperative chemotherapy
HER 2 expression | through study completion, an average of 1 year
  To determine the number of patients with HER2 overexpressing gastric cancers

CONTACTS AND LOCATIONS:
Overall Officials: Bettina G Muller, MD, Principal Investigator — Grupo Oncologico Cooperativo Chileno de Investigation
Locations (1):
- Instituto Nacional del Cáncer, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
IPD are planned to be shared once the final results have been published, foreseen for 2018, data include all datapoints incorporated in the anonymized data base. The investigators who wish to use the data should submit the protocol (approved by an IRB) and the request to access the database to GOCCHI (admin@gocchi.org)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: December 2019, for 10 years
Access Criteria: The investigators who wish to use the data should submit the protocol (approved by an IRB) and the request to access the database to GOCCHI (admin@gocchi.org)

REFERENCES:
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Okines AFC, Norman AR, McCloud P, Kang YK, Cunningham D. Meta-analysis of the REAL-2 and ML17032 trials: evaluating capecitabine-based combination chemotherapy and infused 5-fluorouracil-based combination chemotherapy for the treatment of advanced oesophago-gastric cancer. Ann Oncol. 2009 Sep;20(9):1529-1534. doi: 10.1093/annonc/mdp047. Epub 2009 May 27. PMID 19474114
- [Background] Garcia CC, Benavides CC, Apablaza SP, Rubilar PO, Covacevich SR, Penaloza PM, Guerra JC, Horwitz BZ, Domancic PH, Bustamante R M, Romero S C. [Surgical treatment of gastric cancer: results in 423 cases]. Rev Med Chil. 2007 Jun;135(6):687-95. Epub 2007 Aug 22. Spanish. PMID 17728893
- See also: Homepage of the Chilean Cooperative Group for Oncological Research — http://www.gocchi.org